CLINICAL TRIAL: NCT00000850
Title: The Effects of GM-CSF on Plasma HIV-1 RNA and Chemokine Receptor Expression in HIV-1 Infected Subjects Receiving Concomitant Potent Antiretroviral Therapy
Brief Title: The Effectiveness of GM-CSF in HIV-Positive Patients Who Are Also Receiving Anti-HIV Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5041; AACTG A5041; 10887 (Registry Identifier: DAIDS ES Registry Number); ACTG A5041 (Other: ACTG)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Granulocyte-Macrophage Colony-Stimulating Factor; RNA, Viral; Anti-HIV Agents; Viral Load; Receptors, Chemokine
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; sargramostim

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Sargramostim

SUMMARY:
The purpose of this study is to see how HIV-positive patients who are taking anti-HIV drugs and have a viral load (level of HIV in the blood) of 1,500 copies/ml or more respond to GM-CSF (granulocyte-macrophage colony-stimulating factor).

GM-CSF is a medication that is being tested in HIV-positive patients to see if it can improve their immune systems or if it can lower the level of HIV in their blood. GM-CSF is often given to patients with leukemia or patients who have received bone marrow transplants to increase their white blood cells and to improve their immune systems. Doctors believe that GM-CSF can increase CD4 counts in HIV-positive patients, but this study will also look at how GM-CSF affects viral load.

DETAILED DESCRIPTION:
GM-CSF promotes the differentiation and activation of granulocytes, monocytes, macrophages, and dendritic cells and enhances the function of these cells. The various cellular responses (i.e., division, maturation, activation) are induced when GM-CSF binds to specific receptors expressed on the surface of target cells. At higher doses, such as the dose used in this protocol, GM-CSF may result in a rapid rise in white blood cell count. However, further research is necessary to determine the potential antiviral effect of GM-CSF in a potent ART-treated population. It is hoped that GM-CSF can decrease the extent of ongoing HIV replication via alteration of macrophage activation and chemokine receptor expression and that this effect can result in reduction of the pool of latently infected T cells.

Patients are stratified at study entry according to screening CD4 count (below 200 cells/mm3 versus 200 cells/mm3 or higher) and screening HIV-1 RNA copy number (between 1,500 and 10,000 versus 10,000 copies/ml or higher). Then, patients are randomized to receive GM-CSF or GM-CSF placebo subcutaneously 3 times per week for 16 weeks. All patients remain on their current stable potent ART (not provided by this study). During Step 2, all patients receive open-label study treatment, consisting of current potent ART plus GM-CSF subcutaneously 3 times per week for 32 additional weeks. HIV-1 RNA, CD4 counts, and clinical and safety parameters are monitored for all patients periodically until Week 52. Patients who experience an increase in HIV-1 RNA of greater than 1 log 10 from baseline on 2 consecutive determinations or a greater than 50% decrease in CD4 count from baseline (a drop of at least 50 cells) on 2 consecutive determinations at any time during Step 1 or 2 must discontinue all study treatment. Patients who discontinue study treatment for any reason prior to Week 16 continue following the study visit schedule through Week 16.

Additional laboratory samples are performed on patients participating in the immunology substudy (ACTG A5042s) in order to further evaluate the effects of GM-CSF on immune function.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a stable viral load of at least 1,500 copies/ml within 30 days of study entry.
* Are on stable aggressive anti-HIV therapy for at least 8 weeks before study entry and intend to remain on this therapy during the study.
* Agree to learn how to give themselves the GM-CSF shots.
* Agree to practice acceptable barrier methods of birth control (such as condoms) during the study and for at least 12 weeks after treatment ends.
* Are at least 18 years old.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an infection or other illness within 14 days of study entry.
* Have certain types of hepatitis within 30 days of study entry.
* Have a fever or chronic diarrhea within 30 days of study entry.
* Have cancer (except for certain types of Kaposi's sarcoma).
* Have heart disease.
* Are allergic to GM-CSF.
* Have received certain medications.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jacobson, Study Chair; Gail Skowron, Study Chair; Pablo Tebas, Study Chair; Hernan Valdez, Study Chair
Locations (39):
- United States (39):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente LAMC, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - Marin County Specialty Clinic, San Rafael, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington